CLINICAL TRIAL: NCT04149145
Title: Trial of M4344 and Niraparib in Patients With PARP Resistant Recurrent Ovarian Cancer
Brief Title: Trial of M4344 and Niraparib in Patients With Poly (ADP-ribose) Polymerase (PARP) Resistant Recurrent Ovarian Cancer
Acronym: PARP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: never opened
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rebecca Arend, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB1885
Record Dates: First submitted 2019-10-23; First posted 2019-11-04 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer Recurrent
Keywords: Ovarian Cancer; PARP Resistant; ATR inhibitor; M4344; Niraparib
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M4344+Niraparib (Experimental): all PARP resistant, recurrent ovarian cancer
  Interventions: Drug: M4344+Niraparib

INTERVENTIONS:
Drug: M4344+Niraparib — The first phase will be a 3+3 design of fixed dose Niraparib by mouth (PO) every day (QD) and M4344 will be escalated from 100-200 mg PO QD (28-day cycle). There will be a 4-week lead in with niraparib only.
  Other Names: PARPi+ATRi
Drug: M4344+Niraparib — In the second phase eligible patients will receive combination Niraparib + the determined dose of M4344 from the first phase.
  Other Names: PARPi+ATRi

SUMMARY:
The purpose of this study is to find out if a new drug, M4344, is safe and has beneficial effects when given in combination with the PARP inhibitor, Niraparib, in women with recurrent ovarian cancer that has progressed while on a PARP inhibitor.

DETAILED DESCRIPTION:
The primary, secondary, and exploratory objective are to assess the safety of the combination of M4344 and Niraparib in a phase 1 trial of patients with PARP resistant recurrent ovarian cancer; to determine the response rate and percentage of participants who remain progression free survival (PFS) at 6 months (%PFS) among ovarian cancer participants that have become resistant to poly (adenosine diphosphate [ADP]) ribose polymerase inhibitors (PARPi) who are treated with ataxia telangiectasia and Rad3-related protein inhibitors (ATRi) + Niraparib in the dose expansion cohort; and to identify potential biological predictors of response and progression of disease with the combination of M4344 and Niraparib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with advanced epithelial serous ovarian cancer, primary peritoneal cancer or fallopian tube cancer
* Patients must have PARP resistant ovarian cancer, defined as progression while being treated with a PARP inhibitor.
* Patients must have at least one lesion that meets the definition of measurable disease by RECIST v1.1.
* Patients must have received at least one but no more than five prior systemic treatment regimens
* Female patients ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Patients cannot have had primary platinum refractory cancer, i.e. documented cancer progression while receiving platinum or within one month of receipt of a platinum based regimen.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment. In addition, patients cannot have been diagnosed with another malignancy within 3 years of starting treatment. Exceptions include fully resected basal cell carcinoma of the skin or squamous cell carcinoma of the skin, in situ cervical cancer, fully resected ductal carcinoma in situ, and stage IA, noninvasive grade I endometrioid endometrial cancer, that has undergone curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include clinically active and significant carcinomatous meningitis that is excluded regardless of clinical stability.
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with treatment emergent adverse events as defined by CTCAE v.4.03 | Baseline through 1 year
  Number and percentage of patients with treatment emergent adverse events and toxicity based upon CTCAE v.4.03 scoring.
Maximum tolerated dose (MTD) of M4344 and Niraparib as defined by CTCAE 4.03 | Baseline through 1 year
  To determine the MTD of M4344 and Niraparib during the dose escalation as defined by CTCAE v.4.03

SECONDARY OUTCOMES:
Overall Response Rate (ORR) as defined by RECIST v.1.1 | Baseline through 6 months
  To determine response rate among ovarian cancer patients that have become resistant to PARPi who are treated with ATRi + Niraparib as defined by RECIST v.1.1.
Percentage progression free survival (PFS) as defined by RECIST v.1.1 | Baseline through 6 months
  To determine percentage of patients who remain progression free at 6 months (%PFS) among ovarian cancer patients that have become resistant to PARPi who are treated with ATRi + Niraparib as defined by RECIST v.1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Arend, MD, MSPH, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
To-Be-Determined

REFERENCES:
- [Derived] Jo U, Senatorov IS, Zimmermann A, Saha LK, Murai Y, Kim SH, Rajapakse VN, Elloumi F, Takahashi N, Schultz CW, Thomas A, Zenke FT, Pommier Y. Novel and Highly Potent ATR Inhibitor M4344 Kills Cancer Cells With Replication Stress, and Enhances the Chemotherapeutic Activity of Widely Used DNA Damaging Agents. Mol Cancer Ther. 2021 Aug;20(8):1431-1441. doi: 10.1158/1535-7163.MCT-20-1026. Epub 2021 May 27. PMID 34045232